CLINICAL TRIAL: NCT01951716
Title: Effects of Xenin-25 on Insulin Secretion and Gastric Emptying in Humans With and Without a Complete Truncal Vagotomy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 08-0861 D
Record Dates: First submitted 2013-09-23; First posted 2013-09-27 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Does the Vagus Nerve Mediate the Effects of Xenin-25
Keywords: Vagotomy; Vagus Nerve; Xenin-25; GIP; Insulin Secretion; Glucagon Secretion; Gastric Emptying
MeSH Terms: interventions — Albumins; xenin 25; monooxyethylene trimethylolpropane tristearate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Truncal Vagotomy (Experimental): Healthy participants without diabetes who have undergone a complete truncal vagotomy
  Interventions: Drug: Graded Glucose Infusion with Placebo; Drug: Graded Glucose Infusion with GIP Alone; Drug: Graded Glucose Infusion with xenin-25 alone; Drug: Graded Glucose Infusion with GIP plus xenin-25; Drug: Meal Tolerance Test with Placebo; Drug: Meal Tolerance Test with xenin-25
- No Vagotomy (Experimental): Healthy participants without diabetes who have not had a complete truncal vagotomy
  Interventions: Drug: Graded Glucose Infusion with Placebo; Drug: Graded Glucose Infusion with GIP Alone; Drug: Graded Glucose Infusion with xenin-25 alone; Drug: Graded Glucose Infusion with GIP plus xenin-25; Drug: Meal Tolerance Test with Placebo; Drug: Meal Tolerance Test with xenin-25

INTERVENTIONS:
Drug: Graded Glucose Infusion with Placebo — Starting at 0 minutes, glucose infusion rates will be increased to 1, 2, 3, 4, 6, and 8 mg/kg/min every 40 minutes.
  Starting at 0 minutes, a primed-continuous intravenous infusion of saline containing 1% human albumin will continue for 240 minutes.
  The study is finished at 240 minutes.
  Other Names: GGI with Albumin Alone
Drug: Graded Glucose Infusion with GIP Alone — Starting at 0 minutes, glucose infusion rates will be increased to 1, 2, 3, 4, 6, and 8 mg/kg/min every 40 minutes.
  Starting at 0 minutes, a primed-continuous intravenous infusion of GIP in saline containing 1% human albumin will continue for 240 minutes.
  The study is finished at 240 minutes.
  Other Names: GGI with GIP
Drug: Graded Glucose Infusion with xenin-25 alone — Starting at 0 minutes, glucose infusion rates will be increased to 1, 2, 3, 4, 6, and 8 mg/kg/min every 40 minutes.
  Starting at 0 minutes, a primed-continuous intravenous infusion of xenin-25 in saline containing 1% human albumin will continue for 240 minutes.
  The study is finished at 240 minutes.
  Other Names: GGI with Xenin
Drug: Graded Glucose Infusion with GIP plus xenin-25 — Starting at 0 minutes, glucose infusion rates will be increased to 1, 2, 3, 4, 6, and 8 mg/kg/min every 40 minutes.
  Starting at 0 minutes, a primed-continuous intravenous infusion of GIP plus xenin-25 in saline containing 1% human albumin will continue for 240 minutes.
  The study is finished at 240 minutes.
  Other Names: GGI with GIP plus Xenin
Drug: Meal Tolerance Test with Placebo — At 0 minutes, a liquid mixed meal (Boost Plus) plus acetaminophen will be ingested.
  Starting at 0 minutes, a primed-continuous intravenous infusion of saline containing 1% human albumin will continue for 300 minutes.
  The study is finished at 300 minutes.
  Other Names: MTT with Albumin Alone
Drug: Meal Tolerance Test with xenin-25 — At 0 minutes, a liquid mixed meal (Boost Plus) plus acetaminophen will be ingested.
  Starting at 0 minutes, a primed-continuous intravenous infusion of xenin-25 in saline containing 1% human albumin will continue for 300 minutes.
  The study is finished at 300 minutes.
  Other Names: MTT with xenin

SUMMARY:
Glucose-dependent Insulinotropic Polypeptide (GIP) and xenin-25 are peptide hormones produced/released from your intestines and help regulate blood sugar levels after you eat. We have previously performed studies in humans that measured the effects of xenin-25 and GIP (alone and together) on blood sugar levels. One study was conducted with an intravenous infusion of glucose but without ingestion of a meal. In this study, xenin-25 increased the effects of GIP on insulin secretion- but only in humans without type 2 diabetes mellitus (T2DM). A second study was conducted in conjunction with ingestion of a meal. In this study, xenin-25 reduced blood glucose levels by delaying gastric emptying and this effect was similar in humans with and without T2DM. A variety of studies that we have performed suggest that xenin-25 works by activating nerves. A specific nerve called the vagus nerve plays an important role in regulating insulin secretion. This study will determine if the vagus nerve (which was disrupted if you had a vagotomy) is needed for the effects of xenin-25 on insulin secretion and/or gastric emptying.

DETAILED DESCRIPTION:
Two groups of subjects, both without T2DM, will be studied. One group will consist of people who previously received a complete truncal vagotomy as part of a surgical treatment unrelated to this research project. The other group will be subjects who have not had a truncal vagotomy.

Initially, each potential participant will be administered an oral glucose tolerance test at the screening visit to make sure that they do not have type 2 diabetes. They will also have a sham feeding test to check for the completeness (or absence) of the vagotomy. As outlined below, each subject will then receive 4 graded glucose infusions (GGI) and 2 meal tolerance tests (MTT)- each on a separate occasion following an overnight fast.

For each GGI, the subject will be given an intravenous infusion of glucose such that blood glucose levels slowly increase over a 4 hour period. On separate occasions, the participant will also receive a primed-continuous infusion of GIP alone, xenin-25 alone, GIP plus xenin-25, or placebo (constant dose of 4 pmoles x kg-1 x min-1). Blood samples will be collected before and during the GGI for the measurement of glucose, insulin, C-peptide, glucagon, pancreatic polypeptide, GIP and xenin-25 levels. Insulin secretion rates will also be calculated. By comparing results for the two groups, we will learn if the vagus nerve mediates the effects of GIP, xenin-25, or the combination of GIP plus xenin-25 on insulin secretion in humans and thus, if this signaling circuit is impaired in humans with T2DM.

For the MTTs, the participant will ingest a liquid meal (Boost Plus) plus acetaminophen (Tylenol). On separate occasions, a primed-continuous infusion of vehicle alone or xenin-25 alone (constant dose of 12 pmoles x kg-1 x min-1) will be initiated at the same time the meal is ingested. Blood samples will be collected before and during the MTT for the measurement of acetaminophen, glucose, insulin, C-peptide, glucagon, GIP and xenin-25 levels. Insulin secretion rates will also be calculated. The rate of acetaminophen appearance in the blood is an indirect measure of the rate of gastric emptying. By comparing results for the two groups, we will learn if the vagus nerve mediates the effects of xenin-25 on gastric emptying in humans.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70. No minors will be studied.
* Individuals must be able to consent for their own participation (no mental impairment affecting cognition or willingness to follow study instructions).
* Healthy volunteers with no clinical evidence of Type 2 Diabetes
* Healthy volunteers who have undergone a complete truncal vagotomy
* Healthy volunteers who have not had a complete truncal vagotomy
* Women of childbearing potential must be currently taking/using a method of birth control that is acceptable to the investigators. A pregnancy test will be done at the beginning of each visit. Any woman with a positive pregnancy test will be removed from the study.
* Willingness to complete all required visits

Exclusion Criteria:

* <18years of age or >70 years of age
* Lacks cognitive ability to sign the consent &/or follow the study directions for themselves
* Women unwilling to comply with using an acceptable method of contraception during the course of the study, or who are currently breast-feeding.
* Volunteers with Type 2 diabetes
* Volunteers with a history of Acute Pancreatitis
* Volunteer with a history of Chronic Pancreatitis and/or risk factors for chronic pancreatitis including hypertriglyceridemia (triglycerides >400mg/ml) hypercalcemia (blood calcium level >11.md/dl) and/or the presence of gallstones.
* Volunteers with a history of gastrointestinal disorders, particularly related to gastric motility/emptying such as gastric bypass, documented gastro-paresis in diabetic volunteers.
* Volunteers with a history of cancer. Exception: skin cancer.
* Known heart, kidney. liver or pancreatic disease requiring medications.
* Subjects unwilling to allow the use of their own blood or the human albumin in the preparation of the peptides.
* Unwillingness to allow blood glucose level adjustment (if needed) with IV insulin.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Insulin secretion rates will be measured during the GGI and MTTs | 3 years

SECONDARY OUTCOMES:
Plasma acetaminophen levels will be measured during MTTs | 3 years

OTHER OUTCOMES:
Plasma glucose levels will be measured during the GGIs and MTTs. | 3 years
Plasma glucagon levels will be measured during the GGIs and MTTs. | 3 years
Plasma insulin levels will be measured during the GGIs and MTTs. | 3 years
Plasma C-peptide levels will be measured during the GGIs and MTTs. | 3 years
Plasma pancreatic polypeptide levels will be measured during the GGIs and MTTs. | 3 years
Plasma GIP levels will be measured during the GGIs and MTTs. | 3 years
Plasma xenin-25 levels will be measured during the GGIs and MTTs. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Burton M Wice, PhD, Principal Investigator — Washington University School of Medicine; Dominic Reeds, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States